CLINICAL TRIAL: NCT07086508
Title: A Randomized Clinical Trial: Examining the Efficacy of eCHECKUP TO GO Combined With a Brief Parent-based Intervention to Reduce High School Student Drinking
Brief Title: Examining an Intervention to Reduce High School Drinking
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Binghamton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00006200
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Underage Drinking; Drinking, Teen; Adolescent Alcohol Use
Keywords: Underage drinking; Teen Alcohol Use
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Intervention Model Description: The first group receives the e-CTG and the second group receives the e-CTG+.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-CHECKUP TO GO (eCTG) (Experimental): A brief, web-based program designed by San Diego State University to reduce high-risk drinking by providing personalized normative feedback regarding alcohol use, risk factors, and risks associated with drinking and accurate information about alcohol
  Interventions: Behavioral: e-CHECKUP TO GO (eCTG)
- e-Parent Intervention and eCTG (eCTG+) (Experimental): The eCTG+ is a combination of the eCTG and the e-Parent Intervention, which is an electronic handbook developed by Rob Turrisi to guide parents in discussing drinking, behaviors, and consequences with their teens.
  Interventions: Behavioral: e-Parent Intervention and eCTG (eCTG+)

INTERVENTIONS:
Behavioral: e-CHECKUP TO GO (eCTG) — A brief, web-based program designed by San Diego State University to reduce high-risk drinking by providing personalized normative feedback regarding alcohol use, risk factors, and risks associated with drinking and accurate information about alcohol.
  Arms: e-CHECKUP TO GO (eCTG)
Behavioral: e-Parent Intervention and eCTG (eCTG+) — The eCTG+ is a combination of the eCTG and the e-Parent Intervention, which is an electronic handbook developed by Rob Turrisi to guide parents in discussing drinking, behaviors, and consequences with their teens.
  Arms: e-Parent Intervention and eCTG (eCTG+)

SUMMARY:
Underage drinking is a significant problem in the United States. While past research supports the efficacy of interventions in delaying the initiation of alcohol use implemented in middle school and early high school, research shows drinking by older high schoolers is problematic and interventions for older high schoolers remain limited. The current project will test the efficacy of the e-CHECKUP TO GO (eCTG), alone and combined with an electronic-Parent-Based Intervention (ePBI), for junior and senior high school students using a nationally representative sample with the goal of reducing alcohol use and negative consequences.

DETAILED DESCRIPTION:
Prevalence rates of high school alcohol use suggest 61.6% of high school students have used alcohol by their senior year and 1 in 3 students report alcohol use past 30-days. High school risky drinking is associated with negative consequences including impaired neurocognitive functioning, academic problems, hangovers, passing out, unwanted sex, dating violence, suicide attempts, illicit drug use, riding with impaired drivers, and impaired driving.

While past research supports the efficacy of interventions in delaying the initiation of alcohol use implemented in middle school and early high school, research shows drinking by older high schoolers is problematic and interventions for older high schoolers remain limited. Implementation with high schoolers has always been difficult to sustain following the completion of the grant funding period due to large costs associated with personnel to hire, train, and supervise teachers and staff to implement interventions with fidelity. As an alternative, brief web-based personalized feedback interventions that do not require staffing or costs to implement to large numbers of students have shown promise (e.g., eCHECKUP TO GO; eCTG). Our preliminary work, including our funded NIAAA R21 study, supporting this proposal has shown eCTG is efficacious in changing normative perceptions of peer drinking frequency and drunkenness, positive alcohol expectancies, and reducing both alcohol use and consequences among high school students. The proposed research will expand on these findings by conducting a randomized controlled trial using the eCHECKUP TO GO (eCTG) alone and combined with an efficacious brief electronic-Parent-Based Intervention on a nationally representative sample of high school juniors and seniors.

The design is a two-arm RCT: eCTG and eCTG+. Data collection will occur across 5 waves (pre-intervention baseline, 1-, 3-, 6-, and 9- month follow-ups) for the three intervention arms. In all arms there is one wave for parents (baseline only)

ELIGIBILITY:
Inclusion Criteria:

* Teen is aged 15-18/Parent has a teen aged 15-18
* Parent and teen both consent (forming a dyad testing unit)
* They are part of Ipsos' Knowledge Panel

Exclusion Criteria:

* Outside of the teen age range/Parent does not have a teen aged 15-18

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Examine changes in alcohol use | Baseline, 3 month, 6 month, 9 month, 12 month
  A standard drink definition will be provided, indicating that a standard drink consists of 12 oz. of beer or wine cooler, 8.5 oz. of malt liquor, 4 oz. of wine, or 1.5 oz. of hard liquor. Using the Timeline Followback (TLFB; Sobell & Sobell, 1996) participants will indicate how many drinks they consumed on each day of the past three months. For days alcohol was consumed, participants will also note the number of hours spent drinking.

SECONDARY OUTCOMES:
Examine Changes in Consequences of Alcohol Use | Baseline, 3 month, 6 month, 9 month, 12 month
  Alcohol-related consequences (e.g., said or done embarrassing things, blackout) from the past three months will be measured using the established Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ; Read, Kahler, Strong, & Colder, 2006). Response options will be measured on a 7-point scale ranging from (0) no, not in the past year to (6) 11 or more times in the past three months.

OTHER OUTCOMES:
Examine Changes in Parental Rules about Underage Drinking (Permissiveness) | Baseline, 3 month, 6 month, 9 month, 12 month
  Adapted from measures by Van Der Vorst et al. (2006), parental permissiveness of underage drinking will be assessed using six items (e.g., I am allowed to drink alcohol on special occasions), based on level of agreement on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Parental Communication | Baseline, 3 month, 6 month, 9 month, 12 month
  Parental communication about alcohol use will be assessed separately for mothers and fathers. Participants will be asked whether their parent discussed these topics (yes/no) with them within the past three months. Items include topics such as "the importance of not being pressured to drink to fit it".
Examine Changes in Parental Communications | Baseline, 3 month, 6 month, 9 month, 12 month
  General Communication (e.g., my mother/father is there for me when I want to talk) will be assessed separately for mothers and fathers based on level of agreement on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in General Parental Practices | Baseline, 3 month, 6 month, 9 month, 12 month
  General Parenting Practices (e.g., if I had a personal problem I could ask my mother/father for help) will be assessed separately for mothers and fathers based on level of agreement on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Parental Monitoring | Baseline, 3 month, 6 month, 9 month, 12 month
  Parental monitoring (e.g., my mother/father tries to know about my drinking) will be assessed separately for mothers and fathers based on level of agreement on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Alcohol Use Motives | Baseline, 3 month, 6 month, 9 month, 12 month
  Motives will be assessed for using alcohol (e.g., to be sociable; Cooper, 1994). Responses will be recorded using 5-point scale ranging from (1) almost never/never to (5) almost always/always.
Examine Changes in Alcohol Use Expectancies | Baseline, 3 month, 6 month, 9 month, 12 month
  Expectancies for using alcohol (e.g., I will feel badly about myself because of my drinking) will be measured. Responses will be recorded using 7-point scale ranging from (1) strongly disagree to (7) strongly agree.
Examine Changes in Peer Descriptive Norms | Baseline, 3 month, 6 month, 9 month, 12 month
  Perceived peer descriptive norms of drinking will be measured using the Daily Drinking Questionnaire (DDQ; Collins, Parks, & Marlatt, 1985) by assessing how much alcohol, on average, participants' closest friends drink each day of the week.
Examine Changes in Peer Injunctive Norms | Baseline, 3 month, 6 month, 9 month, 12 month
  Perceived peer injunctive norms will be measured by indicating the level of approval participants' closest friends would have from a list of items (e.g., drinking alcohol every weekend) on a 7-point scale ranging from (1) strongly disapprove to (7) strongly approve.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Mastroleo, PhD, Principal Investigator — Binghamton University
Locations (1):
- Binghamton University, Binghamton, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of funding requirements, data collected will be submitted to the NIAAA Data Archive.
Access Criteria: Individuals will request access to the data via a data access request through the data archive.